CLINICAL TRIAL: NCT03157531
Title: Safety and Effectiveness Evaluation of Eximo Medical's B-Laser™ Atherectomy Device, in Subjects Affected With Infrainguinal PAD
Brief Title: Safety and Effectiveness of B-Laser™ in Subjects Affected With Infrainguinal PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eximo Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX-PAD-03
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-05

CONDITIONS: PAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- B-Laser™ Atherectomy System (Experimental): B-Laser™ Atherectomy System
  Interventions: Device: B-Laser™ Atherectomy System

INTERVENTIONS:
Device: B-Laser™ Atherectomy System — The B-Laser™ is indicated for use for atherectomy of infrainguinal stenoses

SUMMARY:
This is a prospective, single-arm, multi-center, international, open-label, clinical study.

DETAILED DESCRIPTION:
The aim of the study is to assess the safety and efficacy of the Eximo Medical's B-Laser™ Atherectomy catheter in subjects with infrainguinal Peripheral Artery Disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. Subject is a candidate for atherectomy for infrainguinal peripheral artery disease.
3. Documented symptomatic atherosclerotic peripheral artery disease Rutherford Classification 2-4.
4. Subject has an infrainguinal target lesion(s) with any type of stenosis (naïve recurrent, or in-stent) estimated to be ≥70% based on CT angiogram or any other imaging modality.
5. Subject is capable and willing to comply with the scheduled follow up
6. Subject or appropriate legal surrogate is able and willing to sign a written Informed Consent Form (ICF).

Intraoperative inclusion criteria (by fluoroscopy angiogram):

1. Target lesion has a stenosis estimated to be ≥70%.
2. In ATK subjects - at least one patent tibial run-off vessel into the foot

   -

Exclusion Criteria:

1. Target lesion is in a vessel graft or synthetic graft.
2. Target lesion length <1cm and >15 cm (in ISR cases could be >25cm).
3. Endovascular or surgical procedure in the target limb performed less than or equal to 30 days prior to the index procedure OR Planned endovascular or surgical procedure 30 days after the index procedure.
4. Intent to use other atherectomy device in the same procedure.
5. Evidence or history of intracranial or gastrointestinal bleeding, intracranial aneurysm, myocardial infarction or stroke within the past 2 months.
6. Evidence or history of aneurysm in the target vessel within the past 2 months.
7. History of bleeding diathesis, coagulopathy or inability to accept blood transfusions.
8. History of heparin-induced thrombocytopenia (HIT) or inability to tolerate antiplatelet medication(s), anticoagulation, or thrombolytic therapy.
9. Subjects requiring dialysis.
10. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
11. Serious illness that may affect subject compliance to protocol and 30-day follow-up.
12. Participating in another clinical study
13. Subject is pregnant or planning to become pregnant during the study period.
14. Life expectancy < 12 months
15. Any planned amputation above the ankle.

Intraoperative exclusion criteria (by fluoroscopy angiogram):

1. Inability to intraluminally cross and secure a 0.014" wire across the target lesion.
2. Target lesion length <1cm and >15 cm (in ISR cases >25cm).
3. Reference vessel lumen diameter proximal to target lesion is <150% of the outer diameter of the B-LaserTM.
4. Any clinical and/or angiographic complication prior to the planed insertion of B-laser™.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rundback, Dr., Principal Investigator — Holy Name Medical Center, Teaneck, New Jersey, United States, 07666
Locations (11):
- United States (8):
  - Arkansas Heart, Little Rock, Arkansas
  - Orlando Health, Altamonte Springs, Florida
  - Cardiovascular solutions institute, Blake MC, Bradenton, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - UnityPoint Trinity Bettendorf , Genesis Health System, Davenport, Iowa
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
- Medical University Graz, Graz, Austria
- Italy (2):
  - Policlinico Abano Terme, Abano Terme
  - Maria Cecilia Hospital, Cotignola

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | B-Laser™ Atherectomy System
Started | 97
Analyzed at 30 Days For MAEs | 93
Completed | 91
Not Completed | 6
Not completed — Death | 2
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lesions
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 97
Number analyzed (Lesions) | 107
Age, Continuous [Mean (Full Range); unit: years] | 70.5 [46 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 83
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 13
  United States | 77
  Italy | 7
Rutherford class at baseline [Mean (Standard Deviation); unit: scores on a scale] — Rutherford Classification is determined by the physician and represents the progress of the peripheral artery disease. It has seven stages, from Stage 0 to Stage 6, when the lower value indicates a better outcome: 0= Asymptomatic; 1= Mild claudication; 2= Moderate claudication; 3= Severe claudication; 4= Rest pain; 5= Ischemic ulceration not exceeding ulcer of the digits of the foot; 6= Severe ischemic ulcers or frank gangrene.
  scores on a scale | 2.77 (0.60)
WIQ (Walking Impairment Questionnaire) at baseline [Mean (Standard Deviation); unit: scores on a scale] — WIQ is a patient fulfilled survey reporting the grade of ones physical activities ability to represent the progress of the peripheral artery disease. It has few subscales (walking speed, distance, climbing stairs), when the total score of this survey ranges between 0 (worst) and 100 (best), and the higher value = the better outcome. Population: Unavailable data for 4 participants out of the 97.
  scores on a scale
    number analyzed (Participants) | 93
    (all) | 0.23 (0.22)
ABI (Ankle Brachial Index) at baseline [Mean (Standard Deviation); unit: ratio] — ABI is calculated as the ratio of blood pressure in the ankle to the arm blood pressure. The normal value ranges between 0.9 to 1.3. An index under 0.90 means that blood is having a difficult time getting to the legs and feet: 0.41 to 0.90 indicates mild to moderate peripheral artery disease; 0.40 and lower indicates severe disease. Population: Unavailable data for 9 participants out of the 97.
  ratio
    number analyzed (Participants) | 88
    (all) | 0.71 (0.19)
Baseline Stenosis % at target lesion (by Core laboratory) [Mean (Standard Deviation); unit: %] | 85.7 (12.2)
Baseline Stenosis % at target lesion (by Core laboratory) [Count of Units; unit: Lesions]
  Stenosis ≤ 95% | 72
  Stenosis > 95% and ≤ 99% | 12
  Chronic total occlusion (stenosis 100%) | 23
Baseline Calcification level at target lesion (by Core laboratory) [Count of Units; unit: Lesions]
  no | 24
  mild/moderate | 55
  severe | 28
Target lesion length (by Core laboratory) [Mean (Full Range); unit: cm] | 5.4 [1.0 to 23.7]

OUTCOME MEASURES:

1. Primary Outcome: Acute Technical Success
Description: Reduction from baseline in residual diameter stenosis (%), prior to any adjunctive therapy, achieved by the B-Laser™ catheter
  A change (always a reduction) between two time points (baseline time-point and post B-Laser treatment time-point, both perioperative) is reported:
  * As assessed quantitatively by the core laboratory.
  * This endpoint will be met if the mean reduction in residual diameter stenosis is greater than 20%.
  * A greater reduction means better results.
Time Frame: Perioperative
Population: Unavailable angiographic data for primary efficacy endpoint analysis for 2 participants with 2 lesions out of the 97 participants with 109 lesions (these 2 were considered ITT and not PP).
Measure: Mean (Standard Deviation); unit: Change in RDS (%)
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 95
Number analyzed (lesions) | 107
Change in RDS (%) | 33.6 (14.2)

2. Primary Outcome: Number of Participants With Freedom From 30 Days Major Adverse Events (MAEs)
Description: 1. Unplanned target limb amputation above the ankle
  2. Clinically Driven Target Lesion Revascularization (CDTLR)
  3. Cardiovascular related deaths
     * As adjudicated by the Clinical Event Committee (CEC).
     * This endpoint will be met if the freedom from MAE rate is greater than 85%.
Time Frame: 30 (+/-5) days post procedure
Population: 1 Cardiovascular related death was unrelated to the device per the CEC. Four participants out of the 97 with unavailable data: two were lost to follow-up before the 30-day visit was completed, and two others had their 30-day visit outside of the allowable window (day 16 and day 23).
Measure: Count of Participants; unit: Participants
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 93
Participants | 92

3. Secondary Outcome: Number of Lesions With Freedom From Clinically Significant [1] Device Related Adverse Events (AEs) Requiring Intervention in the Target Vessel
Description: 1. Perforation
  2. Dissection
  3. Distal embolization or in situ thrombus
  4. Pseudoaneurysm
     * As adjudicated by the Clinical Event Committee (CEC). [1] Note: Clinically Significant AEs are defined as adverse events that REQUIRE any intervention,treatment or any hospitalization or its prolongation, in order to prevent death, persistent/significant disability/incapacity or congenital anomaly/birth defect.
Time Frame: Perioperative and up to 30 (+/-5) days post procedure
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 95
Number analyzed (lesions) | 107
lesions | 107

4. Secondary Outcome: Number of Lesions With Freedom From Non-Clinically Significant [1] Device Related Adverse Events (AEs) in the Target Vessel
Description: 1. Perforation
  2. Dissection
  3. Distal embolization or in situ thrombus
  4. Pseudoaneurysm
     * As adjudicated by the Clinical Event Committee (CEC). [1] Note: non-Clinically Significant AEs are defined as adverse events that DO NOT REQUIRE any intervention, treatment or any hospitalization or its prolongation, in order to prevent death, persistent/significant disability/incapacity or congenital anomaly/birth defect.
Time Frame: Perioperative and up to 30 (+/-5) days post procedure
Population: All the 16 cases were type A (11) and B (5) dissections only. No perforations, major dissections, emboli or pseudoaneurysm.
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 95
Number analyzed (lesions) | 107
lesions | 91

5. Secondary Outcome: Number of Lesions With Residual Stenosis by Angiography of ≤ 30% Post-procedure Including Any Adjunctive Therapy, With no Flow Limiting Dissection.
Description: Number of Lesions with residual stenosis by angiography of ≤ 30% post-procedure including any adjunctive therapy, with no flow limiting dissection.
  * As assessed quantitatively by the core laboratory.
Time Frame: Perioperative
Population: Unavailable data for primary efficacy endpoint analysis for 2 participants out of the 97.
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 95
Number analyzed (lesions) | 107
lesions
  Yes | 95
  No | 12

6. Secondary Outcome: PAD Measurements at the 30-day Visit Post-procedure Compared to Baseline (1)
Description: 1. Rutherford Classification: a doctor determined 7 stages scale (0= Asymptomatic, 6= Severe ischemic ulcers/frank gangrene) representing PAD progress, lower value = better outcome. Positive difference between time-points represents a clinical deterioration through time and vice versa.
  2. Walking Impairment Questionnaire (WIQ): a patient fulfilled survey to grade physical ability representing PAD progress, has 3 sub-scales (walking speed, distance, climbing stairs), when the total score ranges between 0-100, higher value = better outcome. Positive difference between time-points represents a clinical improvement through time and vice versa.
Time Frame: 30 (+/-5) days post procedure
Population: Only available data for comparison at the two time-points is presented for each parameter .
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 94
scores on a scale
  Rutherford difference (30 day post-procedure - BL) | -1.79 (1.22)
  WIQ difference (30 day post-procedure - BL): number analyzed (Participants) | 81
  WIQ difference (30 day post-procedure - BL) | 0.26 (0.28)

7. Secondary Outcome: PAD Measurements at the 30-day Visit Post-procedure Compared to Baseline (2)
Description: c) Ankle-Brachial Index (ABI): ankle/arm blood pressure ratio. Normal value ranges between 0.9-1.3. Under 0.9 index means blood has a difficult time getting to legs & feet; 0.4-0.9 indicates mild-moderate PAD; 0.4 and lower indicates severe PAD. Positive difference between time-points represents a clinical improvement through time and vice versa.
Time Frame: 30 (+/-5) days post procedure
Population: Only available data for comparison at the two time-points is presented for each parameter .
Measure: Mean (Standard Error); unit: ratio
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 82
ratio | 0.24 (0.18)

8. Secondary Outcome: Number of Lesions With Clinical Success at 30 Days
Description: Defined as < 50% stenosis at the treated lesion, as assessed quantitatively by duplex ultrasound when the peak systolic velocity ratio is < 2.5.
  * As assessed quantitatively by the core laboratory.
Time Frame: 30 (+/-5) days post procedure
Population: Unavailable PSVR for 13 participants (14 lesions) from 95 participants (107 lesions): 5 participants (6 lesions) not diagnostic due to technical incompliance at exam; 3 participants (3 lesions) lost to follow-up; 1 participant (1 lesion) died; 4 participants (4 lesions), core lab could not calculate PSVR, yet were considered patent by absolute PSV.
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 82
Number analyzed (lesions) | 93
lesions | 90

9. Post Hoc Outcome: Number of Participants With Freedom From 6 Months Major Adverse Events (MAEs) [Not a Study Pre-specified Endpoint]
Description: 1. Unplanned target limb amputation above the ankle
  2. Clinically Driven Target Lesion Revascularization (CDTLR)
  3. Cardiovascular related deaths
     * As adjudicated by the Clinical Event Committee (CEC).
Time Frame: 6 months (+/-14 days) post procedure
Population: 3 CD-TLRs were possibly related to device & definitely related to index procedure, per CEC. 8 participants out of total 97 with unavailable data: 3 subjects were lost to follow-up before 6-month visit was completed, 1 subject died before 6-month visit, and 3 other subjects had their 6-month visit outside of the allowable window (before Day 166).
Measure: Count of Participants; unit: Participants
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 89
Participants | 86

10. Post Hoc Outcome: PAD Measurements at the 6-month Visit Post-procedure Compared to Baseline [Not a Study Pre-specified Endpoint] (1)
Description: as for outcome 6
Time Frame: 6-month (+/-14 days) post-procedure
Population: Only available data for comparison at the two time-points is presented for each parameter .
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 88
score on a scale
  Rutherford difference (6 month post-procedure -BL) | -2.02 (1.12)
  WIQ difference (6 month post-procedure -BL): number analyzed (Participants) | 82
  WIQ difference (6 month post-procedure -BL) | 0.25 (0.30)

11. Post Hoc Outcome: PAD Measurements at the 6-month Visit Post-procedure Compared to Baseline [Not a Study Pre-specified Endpoint] (2)
Description: as for outcome 7
Time Frame: 6-month (+/-14 days) post-procedure
Population: Only available data for comparison at the two time-points is presented for each parameter .
Measure: Mean (Standard Error); unit: ratio
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 79
ratio | 0.17 (0.28)

12. Post Hoc Outcome: Number of Lesions With 6-Month Patency [Not a Study Pre-specified Endpoint]
Description: Defined as < 50% stenosis at the treated lesion, as assessed quantitatively by duplex ultrasound when the peak systolic velocity ratio is < 2.5.
  * As assessed quantitatively by the core laboratory.
  This is not a study pre-specified endpoint.
Time Frame: 6 months (+/-14 days) post procedure
Population: Unavailable PSVR for 14 participants (17 lesions) from 95 participants (107 lesions): 3 participants (4 lesions) not diagnostic due to technical incompliance at exam; 5 participants (5 lesions) lost to follow-up; 2 participants (3 lesions) died; 4 participants (5 lesions), core lab could not calculate PSVR.
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy System
Number analyzed (Participants) | 82
Number analyzed (lesions) | 90
lesions | 77

ADVERSE EVENTS:
Time Frame: 6 months (+/-14 days) post procedure
Description: * All-Cause Mortality: 2 deaths were unrelated to the device, per the CEC
  * Serious Adverse Events: 40/43 SAEs were unrelated to the device. Only 3 'Vascular disorders' SAEs were classified by CEC as 'possibly related' to device and 'definitely related' to procedure (all 3 were CDTLRs).
  * Other (Not Including Serious) Adverse Events: 53/55 AEs were unrelated to the device. Only 2 'Vascular disorders' AEs were classified by CEC as 'possibly related' to device and 'definitely related' to procedure.
Arm/Group | B-Laser™ Atherectomy System
All-Cause Mortality (participants affected / at risk) | 2/93
Serious Adverse Events (participants affected / at risk) | 43/93
Other Adverse Events (participants affected / at risk) | 54/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-Laser™ Atherectomy System (N=93)
General disorders (General disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3)
Renal and urinary disorders (Renal and urinary disorders) | 3 (3)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 4 (4)
Cardiac disorders (Cardiac disorders) | 13 (13)
Vascular disorders (Vascular disorders) | 13 (13)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-Laser™ Atherectomy System (N=93)
Eye disorders (Eye disorders) | 1 (1)
General disorders (General disorders) | 9 (9)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac disorders (Cardiac disorders) | 4 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4 (4)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 9 (9)
Vascular disorders (Vascular disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT03157531/Prot_SAP_000.pdf